CLINICAL TRIAL: NCT02805374
Title: ASP1517 Pharmacokinetic Study - Evaluation of Food Effect on the Pharmacokinetics of ASP1517
Brief Title: A Food Effect Study to Evaluate the Pharmacokinetics of ASP1517
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1517-CL-0202
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; ASP1517; Food effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP1517 fasting then fed (Experimental): Subjects will receive a single oral dose of ASP1517 under fasting conditions in period 1, then subjects will receive a single oral dose of ASP1517 under fed conditions in period 2.
  Interventions: Drug: ASP1517
- ASP1517 fed then fasting (Experimental): Subjects will receive a single oral dose of ASP1517 under fed conditions in period 1, then subjects will receive a single oral dose of ASP1517 under fasting conditions in period 2.
  Interventions: Drug: ASP1517

INTERVENTIONS:
Drug: ASP1517 — Oral

SUMMARY:
The objective of this study is to evaluate the effect of food on the pharmacokinetics of a single oral dose of ASP1517 in non-elderly healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: ≥50.0 kg and <80.0 kg
* Body-mass index : ≥17.6 and <26.4 kg/m2
* Subject must agree to use two of the established contraceptive methods after informed consent acquisition through 84 days after the last administration of the study drug.
* Subject must agree not to donate sperm after informed consent acquisition through 84 days after the last administration of the study drug.

Exclusion Criteria:

* Received or is scheduled to receive any investigational drugs in other clinical trials or post-marketing studies within 120 days before screening or during the period from screening to the hospital admission day of Period 1
* Received or is scheduled to receive medications (including over-the-counter [OTC] drugs) within 7 days before the hospital admission day of Period 1
* Received or is scheduled to receive supplements within 7 days before the hospital admission day of the Period 1
* Deviates from any of the normal range of blood pressure, pulse rate, body temperature and standard 12-lead electrocardiogram (ECG) at screening or the hospital admission day of Period 1
* Meets any of the criteria for laboratory tests at screening or the hospital admission day of Period 1. Normal ranges of each test specified at the test/assay organization will be used as the normal ranges in this study.
* Concurrent or previous drug allergies.
* Development of (an) upper gastrointestinal symptom(s) within seven days before the hospital admission day of Period 1.
* Concurrent or previous hepatic disease, heart disease, respiratory disease, gastrointestinal disease, renal disease, endocrine disease, cerebrovascular disorder, malignant tumor, retinal neovascular lesions and macular edema.
* A history of digestive tract excision.
* Previous use of hypoxia inducible factor-prolyl hydroxylase inhibitors (HIF-PHI) such as ASP1517 (FG-4592), YM311(FG-2216) or erythropoietin products.
* Excessive alcohol or smoking habit.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameter of ASP1517 in Plasma: AUCinf | Up to Day 4 of each treatment period
  AUCinf: Area under the concentration-time curve from the time of dosing extrapolated to time infinity
PK parameter of ASP1517 in Plasma: Cmax | Up to Day 4 of each treatment period
  Cmax: Maximum concentration

SECONDARY OUTCOMES:
PK parameter of ASP1517 in Plasma: AUClast | Up to Day 4 of each treatment period
  AUClast: Area under the concentration-time curve from the time of dosing to the last measurable concentration
PK parameter of ASP1517 in Plasma: CL/F | Up to Day 4 of each treatment period
  CL/F: Apparent total systemic clearance
PK parameter of ASP1517 in Plasma: λz | Up to Day 4 of each treatment period
  λz: Terminal rate constant
PK parameter of ASP1517 in Plasma: MRTinf | Up to Day 4 of each treatment period
  MRTinf: Mean residence time extrapolated to infinity
PK parameter of ASP1517 in Plasma: t1/2 | Up to Day 4 of each treatment period
  t1/2: Terminal elimination half-life
PK parameter of ASP1517 in Plasma: tmax | Up to Day 4 of each treatment period
  tmax: Time of Cmax
PK parameter of ASP1517 in Plasma: tlag | Up to Day 4 of each treatment period
  tlag: Lag time
PK parameter of ASP1517 in Plasma: Vz/F | Up to Day 4 of each treatment period
  Vz/F: Apparent volume of distribution during the terminal elimination phase
PK parameter of ASP1517 in Urine: Ae | Up to Day 4 of each treatment period
  Ae: Cumulative amount of ASP1517 excreted into urine
PK parameter of ASP1517 in Urine: CLR | Up to Day 4 of each treatment period
  CLR: Renal clearance
Safety assessed by adverse events | Up to Day 9 of Period 2
Number of participants with abnormal vital signs and/or adverse events during treatment period | Up to Day 9 of Period 2
Number of participants with abnormal laboratory values and/or adverse events during treatment period | Up to Day 9 of Period 2
Number of participants with abnormal standard 12-Lead ECG and/or adverse events during treatment period | Up to Day 9 of Period 2
  ECG: Electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided